CLINICAL TRIAL: NCT04896411
Title: Choice Of Diction's Effect: Effects in No Code Phrasing on Code Status Discussions
Brief Title: Choice of Diction's Effect
Acronym: CODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Karthik Joshua Kota, MD MPH, Instructor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2020002188
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Communication; Advance Directives; Decision Making; Cardiopulmonary Resuscitation
Keywords: Older Adult; Allow a Natural Death; Do Not Resuscitate; Resuscitation Decisions
MeSH Terms: conditions — Communication | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative Phrase (Experimental): This arm will have the code status question randomized to offer CPR vs the alternative phrase
  Interventions: Other: Alternative phrasing for no code
- Standard of care phrase (Active Comparator): This arm will have the code status question randomized to offer CPR vs the standard of care phrase
  Interventions: Other: Standard of care for no code

INTERVENTIONS:
Other: Alternative phrasing for no code — This intervention will use the alternative phrase noted in the literature when discussing code status. This will be the only intervention, and all other aspects of trial participation will be collection of data
  Arms: Alternative Phrase
Other: Standard of care for no code — This intervention will use the standard of care phrase noted in the literature when discussing code status. This will be the only intervention, and all other aspects of trial participation will be collection of data
  Arms: Standard of care phrase

SUMMARY:
The purpose of the research is to determine how the language used when discussing preferences about cardiopulmonary resuscitation (CPR) affects decisions regarding this (code status)

DETAILED DESCRIPTION:
Most Americans express a preference for dying at home naturally and surrounded by loved ones. However, many also believe that cardiopulmonary resuscitation (CPR) is more effective than it is, and want to have CPR even when the chances for a good outcome is poor. Among other reasons, the alternative term (Do Not Resuscitate, or DNR) has been shown in the literature to be associated by patients with passive, sub-optimal, and low quality care.

This study will attempt to determine patient preference for the "no CPR" term on patients admitted to the hospital using alternate phrasing. During admission to the Medical Teaching Service, patients over the age of 65 who are able to consent and who are not critically ill/unstable will be approached. After checking brief background questions (such as if they ever had discussions like these before), they will be randomized into two groups and asked code status using one of the two phrases. This question will determine the patient's "code status;" asking for this is a routine part of hospitalized care that is required by law (the exact terminology is left to the care team). After determining the patient's code status, they will be asked how satisfied they were with the decision; the investigator will be asked if they agree with the decision separately. Demographic and clinical information will be collected. Six months later, the patient will be contacted again; at this time, they will be asked about recent life and health changes. Finally, they will be asked their code status one more time. This will conclude the participant's involvement in the study

ELIGIBILITY:
Inclusion Criteria:

* 65 or older
* English-fluency in reading and speaking
* Capacity to consent

Exclusion Criteria:

* Unstable psychiatric illness
* Unstable/critically ill patients requiring ICU-level care
* Active substance abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2023-02-08 (Estimated)

PRIMARY OUTCOMES:
Code Status Selection | Immediately collected after consent and randomization into a study arm
  Selection of "code" versus "no code" decision depending on phrasing used, stratified by GO-FAR calculation

SECONDARY OUTCOMES:
Participant Satisfaction with Decision | Immediately collected after consent and randomization into a study arm
  Determine patient satisfaction of, and provider agreement with, code discussion. The former will be measured using a modified Satisfaction with Decision Scale, a six-item Likert scale indicating agreement or not with the statements provided. The latter will be determined by asking the physician if they agree (yes/no/unsure)
Length of Conversation | Immediately collected after consent and randomization into a study arm
  Determine whether there is a difference of conversation length between phrasing groups (measured in minutes)

OTHER OUTCOMES:
Durability of Code Status Decision In the Study Arms at 6 Months (Assessed by Asking Code Status Using the Intervention Phrase Again) | At approximately 6 months, patients will receive a follow-up phone call to determine this
  Determine whether the decision made for code status is durable between the two groups. Patients will again be asked their code status as in outcome 1 during a follow-up phone call (after information about new medical experiences/diagnoses and other code status discussions in the last six months is collected)
Information That May Modify Outcomes 1-4 | Additional information collected "initially" will be at time of consent/randomization into the study arm; additional information collected at "follow-up" will be at approximately six months
  To assess the possibility of other factors modifying the above outcomes, this study will collect additional information. Initially, we will ask about history of prior code status discussion; general demographic information (e.g., income, religion, etc); medical history (including diagnoses, medications, and substance use). At follow-up, we will ask about recent hospitalizations, new medical problems/medications, life stressors (using the Holmes-Rahe Index), and further discussions about code status

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Kota, MD MPH, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared